CLINICAL TRIAL: NCT05181878
Title: AcQMap 2.1 With Electro-Magnetic Tracking System Feasibility Study (EMT Feasibility Study)
Status: Completed | Type: Observational
Sponsor: Acutus Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP-24 US; CLP-24 (EU) (Other: Acutus Medical, Inc.)
Record Dates: First submitted 2021-12-08; First posted 2022-01-06 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Catheter Ablation
Keywords: localization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: The AcQMap 2.1 System with Electro-Magnetic Tracking Feasibility System — Demonstrate the ability of the AcQMap 2.1 System to support EMT in conjunction with the existing impedance localization capabilities. The new EMT technology is expected to continuously provide fully synchronized and similar localization information to the impedance-based localization information associated with the location of the catheter's magnetic sensor position.

SUMMARY:
Non-Significant Risk Clinical Study

Clinical Investigational Use Only for the purposes of collecting electromagnetic tracking data to validate the use of the device in a clinical setting.

DETAILED DESCRIPTION:
The EMT Feasibility Study is a prospective, multi-center, feasibility study designed to demonstrate the feasibility of EMT solution in conjunction with the AcQMap 2.1 System's existing capabilities.

The objective of the study is to demonstrate the ability of the AcQMap 2.1 System to support EMT in conjunction with the existing impedance localization capabilities. The new EMT technology is expected to continuously provide fully synchronized and similar localization information to the impedance-based localization information associated with the location of the catheter's magnetic sensor position.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 years of age or older.
2. Currently scheduled for the ablation of an atrial arrhythmia utilizing the diagnostic AcQMap 2.1 System.
3. Willing and able to give written informed consent.

Exclusion Criteria:

1. In the opinion of the investigator, any contraindication to the planned ablation, including anticoagulation contraindications, atrial thrombus, renal failure, or sepsis.
2. Current enrollment in any study protocol sponsored by Acutus Medical
3. Any other condition that, in the judgment of the investigator, makes the participant a poor candidate for this procedure, the study, or compliance with the protocol (includes vulnerable patient population, mental illness, addictive disease, extensive travel away from the research center, etc.).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any participant 18 years of age or older. Currently scheduled for an ablation of an arrhythmia utilizing the diagnostic AcQMap 2.1 System.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Successful recording of continuous and synchronized impedance and magnetic localization information. | Procedure
  Successful recording of continuous and synchronized impedance and magnetic localization information.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Kansas City Heart Rhythm Institute, Overland Park, Kansas
  - Nevada Heart and Vascular, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: Undecided